CLINICAL TRIAL: NCT01993368
Title: Analysis of Osteoimmune Interactions Linking Inflammation and Bone Destruction in Aggressive Periodontitis
Acronym: PAG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough patient enrolled in the study
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 13-PP-07
Record Dates: First submitted 2013-11-15; First posted 2013-11-25 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Aggressive Periodontitis; Chronic Periodontitis
Keywords: wisdom teeth extraction
MeSH Terms: conditions — Aggressive Periodontitis; Chronic Periodontitis | interventions — Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- chronic periodontitis (Other): biopsy of periodontal granulation tissue (surgical waste)
  Interventions: Other: flow cytometry
- aggressive periodontitis (AP) (Other): biopsy of periodontal granulation tissue (surgical waste)
  Interventions: Other: flow cytometry
- controls (Other): necessitating an extraction of wisdom teeth
  Interventions: Other: flow cytometry

INTERVENTIONS:
Other: flow cytometry — These populations will be identified by different combinations of antibodies to identify:
  * T cell subsets (CD45, CD3, CD4, CD8, CD45RA, CD69, CD28, TCRαβ, TCRγδ, CD197, CD25, FoxP3), B cells (CD45, CD19, HLA-DR, IgA), cells NK (CD45, CD3, CD56).
  * Monocyte subsets (CD45, CD11b, CD14, CD16, CD1c, HLA-DR)
  * Mesenchymal stromal cells (CD45, HLA-ABC, CD105, CD90, CD73)
  Other Names: proportion of lymphocytes, myeloid and mesenchymal populations in the samples, as determined by flow cytometry.

SUMMARY:
Periodontitis are inflammatory diseases characterized by the destruction of the tooth-supporting bone due to increased bone resorption by osteoclasts (OCLs). Two forms are described: chronic periodontitis (CP) and aggressive periodontitis (AP) that differ by the severity and rapidity of bone loss, much more important for AP than CP. In both forms, the link with uncontrolled activation of the immune system is largely admitted. Despite the physiopathology of CP is fairly well studied, very few data are available regarding AP. The investigators aim is to understand the severity of AP by analyzing the proportion and action of immune and mesnchymal cells potentially involved in bone destruction, on biopsies of periodontal granulation tissue (surgical waste) and blood. Three groups of 20 patients will be included: affected with AP, CP or controls (necessitating an extraction of wisdom teeth).

DETAILED DESCRIPTION:
Context: Periodontitis are inflammatory diseases affecting the periodontium and characterized by the destruction of the tooth-supporting bone due to increased bone resorption by osteoclasts (OCLs). Two forms are described: chronic periodontitis (CP) and aggressive periodontitis (AP) that differ by the severity and rapidity of bone loss, much more important for AP than CP. In both forms, the link with uncontrolled activation of the immune system is largely admitted. But despite the physiopathology of CP is fairly well studied, very few data are available regarding AP. Based on the investigators previous studies, their hypothesis to explain this severity is the existence of a vicious circle involving immune cells, mesenchymal cells and OCLs, that would maintain and amplify inflammation and bone loss.

Study: this is a transversal, interventional and single-center study. It includes 3 groups of 20 patients: affected with AP, CP or controls (necessitating an extraction of wisdom teeth).

Aims: the investigators will compare the proportion of immune and mesenchymal cells in the 3 groups of patients to identify the populations potentially involved in bone destruction. The investigators will compare in vitro their capacity to induce OCL differentiation in order to determine their role in bone loss. The investigators will also compare the capacity of OCLs and mesenchymal cells to activate T cells, in order to determine their role in inflammation.

Methodology: patients will be recruited in the department of periodontology, CHU of Nice. After signing the informed consent, a biopsy of periodontal granulation tissue (surgical waste) will be collected during the usual treatment of these diseases, as well as a blood sample. Then, patients will leave the study. Cells from the biopsies will be analyzed by flow cytometry to determine the proportion of lymphocytic, monocytic and mesenchymal cells. In vitro, their capacity to induce OCL differentiation or to activate T cells will be determined. From the blood samples, OCLs will be generated to study their capacity to activate T cells.

Chronology of consultations and examinations: 3 visits are planned: (1) a routine visit corresponding to the usual treatment of the patient during which it is proposed to participate in the study, (2) a visit to obtaining consent, clinical examination, criteria verification and (3) a visit corresponding to the usual treatment in which will be collected tissue biopsies and blood.

ELIGIBILITY:
* Inclusion criterias for agressive periodontits

  * Young patients not suffering of any médical conditions
  * Small amount of calculus detected
  * Pocket depth >5mm
  * Alveolar Bone loss >50%
* Inclusion criterias for chronic periodontitis

  * Evident presence of calculus above or under the gingiva
  * Pocket depth >5mm
* Inclusion criterias for control patients :

  * Young patients in need of impacted wisdom teeth removal
  * And not suffering of chronic or agressive periodontitis
* Exclusion criterias :

  * Patients with blood disorder
  * Patients presenting with liver, kidney, or vascular disorder, and /or psychiatric disorder
  * Patients who have allergies
  * Patients taking biphosphonates, anticoagulant drugs, or anticonvulsivant
  * Patients who have had a cancer of the mouth, and/or treated by radiotherapy
  * Patients who have taken anti-inflammatory drugs, and/or anti-cancer drugs, and/or immuno-suppresive drugs in the past 6 months
  * Patients who have had a periodontal treatment in the past 12 months
  * Pregnant Women
  * Patients juged difficult to follow by the investigator
  * Vulnerable patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
proportion of lymphocytes, myeloid and mesenchymal populations in the samples | At the surgery time
  determined by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme SURMENIAN, MD, Principal Investigator — Odontology Department, NIce University Hospital
Locations (1):
- Odontology Department, Nice Unversity Hospital, Nice, France